CLINICAL TRIAL: NCT02560142
Title: Non-Drug, Single Site, fMRI and Behavior Assessment Optimization Study in Healthy Volunteers
Brief Title: A Non-interventional Functional Magnetic Resonance Imaging (fMRI) Study and Behavioral Assessment in Healthy Participants
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: BP29791
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood for DNA extraction

GROUPS / COHORTS (1):
- All Participants: Healthy participants will undergo behavioral assessment and fMRI.

SUMMARY:
This is a single center non-interventional study in healthy participants for behavioral assessment and fMRI assessments. The study will consist of 2 parts. Part A will involve 5 participants and will study the implementation of the behavioral tests and identify potential issues. Part B will involve 30 participants and will study the test-retest reliability. Duration of participation for each participant will be 30 days for Part A (28 days screening period and 2 days of study visit) and 48 days for Part B (28 days screening period and 2 study visits of 2 days each separated by a period of 14 days).

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants, as determined by screening assessments and principal investigator judgment
* A body mass index (BMI) between 18 to 30 kilogram per square meter (kg/m^2) inclusive with body weight in the range of 50 to 100 kg
* The participant must be able to comply with study requirements as judged by the principal investigator
* Women participants who are not postmenopausal or surgically sterile agree to use effective contraception throughout the study

Exclusion Criteria:

* Female participant with child-bearing potential or a positive blood pregnancy test
* Lactating women participants
* Any history of alcohol and/or drug abuse, addiction or suspicion of regular consumption of drugs of abuse
* Use of any psychoactive medication, or medications known to have effect on central nervous system (CNS) or blood flow
* Any contraindications for magnetic resonance imaging (MRI) scans or any brain/head abnormalities restricting MRI eligibility

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Participants
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Intra Class Coefficient of Correlation (ICC) of the Task Activated Blood Oxygenation Level-Dependent (BOLD) fMRI: Face Matching Task | Day 1
ICC of the Task Activated BOLD fMRI: Monetary Incentive Delay Task | Day 1
ICC of the Task Activated BOLD fMRI: 2 vs 0 Back Working Memory Task | Day 1
ICC of the Task Activated BOLD fMRI: Episodic memory Task (Encoding, Recall, and Recognition of Face-Profession Pairs) | Day 1
ICC of the Task Activated BOLD fMRI: Theory of Mind Task (ToM; To Make Inferences About Others Mental States Using 32 False-Belief Cartoon Stories) | Day 1
ICC of the Resting-State BOLD fMRI, Acquired Using Gradient Echo-Planar Imaging (EPI) Images | Screening (Day -28 to Day -1)
ICC of the Resting-State Arterial Spin Labeling (ASL) to Measure Cerebral Blood Flow, Acquired Using Gradient EPI Images | Screening (Day -28 to Day -1)
ICC of the out of Scanner Behavioral Tasks: Stop Signal Reaction Time (SSRT) to Assess the Time Required to Stop Already Executed Response | Day 1
ICC of the out of Scanner Behavioral Tasks: California Verbal Learning Test - Second Edition (CVLT-II), to Assess an Individual's Episodic Verbal Learning and Memory Abilities | Day 2
Out of Scanner Behavioral Tasks: RAVEN General Intelligence Test | Screening (Day -28 to Day -1)
ICC of the out of Scanner Behavioral Tasks: Emotional Test Battery (ETB), Assessed Using Facial Expression Recognition Task (FERT) and Faces Dot Probe Task (FDOT) to Measure Biases in Emotional Processing | Day 1
ICC of the out of Scanner Behavioral Tasks: Reward Learning Tasks (Reinforcement Learning and Working Memory Task) | Day 2
ICC of the Task Activated BOLD fMRI: Go/No-Go Task | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- PRA Health Sciences Early Development Services, Zuidlaren, Netherlands